CLINICAL TRIAL: NCT03733041
Title: Neuromodulation for Exercise Adherence in Older Veterans
Brief Title: Neuromodulation for Exercise Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2961-R
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Executive Dysfunction; Poor Exercise Adherence
Keywords: exercise adherence; Older veterans; home based exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to parallel groups to receive either the rTMS or sham treatment with allocation ratio of 1:1. The stratified randomization scheme will be generated by a statistician using a random block design with random block sizes, and assignments (X or Y) will be placed in sealed envelopes for sequential opening.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects and the study team (staff responsible for administering treatment or rating outcomes and study physicians) will not know the coil assignment since coils are labeled 'X' or 'Y' and are identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Repetitive Transcranial Magnetic Stimulator (rTMS) treatment and Nintendo Wii-Fit exercises arm (Active Comparator): This group will be randomized to receive Repetitive Transcranial Magnetic Stimulator (rTMS) and Nintendo Wii-Fit exercises
  Interventions: Device: Repetitive Transcranial Magnetic Stimulator; Device: Nintendo Wii-Fit exercises
- Sham treatment and Nintendo Wii-Fit exercises arm (Sham Comparator): This group will be randomized to receive sham treatment and Nintendo Wii-Fit exercises
  Interventions: Device: Sham treatment; Device: Nintendo Wii-Fit exercises
- Nintendo Wii-Fit exercises only arm (Other): This group will not be randomized and receive only Nintendo Wii-Fit exercises
  Interventions: Device: Nintendo Wii-Fit exercises

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulator — Participants randomized to this group will receive repetitive transcranial magnetic stimulation and will do Nintendo Wii-Fit exercises
  Other Names: Nintendo Wii-Fit exercises
  Arms: Repetitive Transcranial Magnetic Stimulator (rTMS) treatment and Nintendo Wii-Fit exercises arm
Device: Sham treatment — Participants randomized to this group will receive sham treatment and will do Nintendo Wii-Fit exercises
  Other Names: Nintendo Wii-Fit exercises
  Arms: Sham treatment and Nintendo Wii-Fit exercises arm
Device: Nintendo Wii-Fit exercises — Participants will do Nintendo Wii-Fit exercises

SUMMARY:
Lack of adherence to an exercise program is a major problem for older Veterans. Several fall prevention programs fail in the home setting due to lack of adherence. Exercise adherence is dependent on brain function among other factors. Magnetic stimulation of the front part of the brain improves brain function necessary for planning and following-through. The investigators propose a three-phase study in 106 sedentary older Veterans. Everyone will be trained on use of the exergames, Nintendo Wii-Fit, that the investigators' team has found beneficial in improving balance and gait. They will be asked to exercise using Wii-Fit at home for 45 minutes daily five days/week for 12-weeks. Those that exercise less than recommended dose and those that exercise adequately but have low executive function will receive either real or sham magnetic stimulation to the front part of their brain over ten sessions paired with exercise training. All subjects will further complete 24-weeks of Wii-Fit home exercises. Adherence, executive function, balance and gait, self-efficacy, delay discounting, and falls will be measured periodically.

DETAILED DESCRIPTION:
Background: Fall-related hospitalizations and consequent morbidity and mortality continue to rise despite the availability for over two decades of evidence-based fall-prevention programs. This is a major problem since more than 2.5 million older adults are treated annually for fall-related injuries in the US. Fall-prevention programs focusing on strength and balance exercises have been successful in facility settings but exercise programs are ineffective at home due to lack of adherence. Estimates indicate that only 1 in 5 individuals adhere to home exercise programs for fall prevention. Thus, there is an urgent need to improve adherence to exercise performed at home by older adults seeking to improve balance for the sake of fall prevention. Behavioral interventions have failed to consistently improve adherence to exercise. Biological reasons for poor exercise adherence, such as executive dysfunction, have not been explored. Adherence to long-term exercise is dependent on executive function (EF), which is controlled by the [dorsolateral prefrontal cortex (DLPFC)] of the brain. EF influences choices in scheduling, forgoing competing activities, enduring subtle costs of time and inconvenience, and the ability to delay gratification. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation increasingly used for neural network specific interventions. rTMS of the DLPFC improves EF, memory, motivation, and mental flexibility. rTMS studies to date have stimulated the motor cortex for gait and balance improvements. The role of DLPFC in exercise adherence has not been explored. The proposed study will be the first to test DLPFC stimulation for improving exercise adherence.

Objective: The study objective is to determine the effects of rTMS treatment of the dorsolateral prefrontal cortex compared to sham on: [1. Short-term (2-wk) changes in executive function;] 2. Long-term (24-wk) adherence to a home-based exercise program; 3. Long-term (24-wk) changes in balance and gait; and [4. Short-term (2-wk) changes in self-efficacy and delay discounting.]

Methods: Sedentary community-dwelling older Veterans (age 60 years and older, [N=106]) will participate in a double-blind randomized sham-controlled three-phase study. The proposed study will use Nintendo Wii-Fit exercises. Phase I will include two weeks of facility-based exercise for safety assessment and learning the program, followed by 12 weeks of home-based exercises. [Subjects with poor adherence and those with good adherence with low EF] will then be randomized to rTMS or sham treatments. Phase II will include ten consecutive weekdays of rTMS or sham treatment along with exercise training for subjects with poor adherence [and for those with good adherence and low EF] and continuation of home-based exercises for those with good adherence and EF. Phase III includes 24-weeks of a home-based exercise program. All subjects will exercise for 45 minutes five days/week. [Objective measure of adherence collected from Wii-Fit console and Conner's continuous performance test for EF will be the primary outcome measures.] Balance and gait will be assessed. [Self-efficacy, delay discounting along with fear of falls, and falls incidence will be assessed. Outcome measures will be assessed at baseline, and at 14, 16, and 40 weeks.]

Significance: This project may have a major impact in improving adherence to an exercise program and in turn, improve balance in sedentary community-dwelling older Veterans. Knowledge gained about the adherence to home-based exercises would be applicable to multiple conditions such as diabetes. Since Wii-Fit and rTMS are readily available, translation of the study results to clinical practice would be expeditious.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary Community Dwelling Veterans age 60 years and older
* Have Television (TV) at home
* Subjects reporting spending long periods of time in sedentary behavior by answering affirmatively to the question: 'For most days, do you feel you sit for too long (6-8 hours or more a day)?

  * Some examples might include when watching TV, working at the computer / laptop or when doing sitting-based hobbies such as reading and sewing' will be included

Exclusion Criteria:

GENERAL EXCLUSION CRITERIA

* Those that participate in regular physical activity for at least 30 minutes five or more days of the week

EXCLUSIONARY DUE TO Wii-Fit Exercises

* Use of wheel chair for mobility
* Cognitive impairment [Montreal Cognitive Assessment (MoCA < 26)]
* Weight 325 lbs. (weight restriction of the Wii-Board)
* Absolute contraindications to exercise per The American College of Sports Medicine guidelines
* Those with medical conditions that in the opinion of the study physician are likely to compromise safe participation

EXCLUSIONARY DUE TO rTMS

* Taking medications known to increase risk of seizures from 2012 Beers criteria such as bupropion, chlorpromazine, clozapine.
* Taking other medications known to increase risk of seizures such as tricyclic antidepressants.
* Taking ototoxic medications: Aminoglycosides, CisplatinHistory of seizures/ seizures in first degree relatives
* Those with implanted device
* History of stroke, aneurysm, or cranial neurosurgery
* History of bipolar disorder
* History of abnormal electroencephalogram (EEG)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Adherence as measured by number of minutes | 14 weeks, 40 weeks
  Total number of minutes exercised
Change in Conner's Continuous Performance Test | 14 weeks, 16 weeks, 40 weeks
  Commission Error percentage Range 0-100% Higher score is improvement
Change in Adherence as measured by number of sessions | 14 weeks, 40 weeks
  Total number of sessions exercised

SECONDARY OUTCOMES:
Change in Gait speed | 14 weeks, 16 weeks, 40 weeks
  The test measures habitual walking speed in meters/sec
Change in Timed Up and Go | 14 weeks, 16 weeks, 40 weeks
  This is a widely accepted test of pro-active balance and mobility and measured in secs

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana P Padala, MD MS, Principal Investigator — Central Arkansas Veterans Healthcare System , Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System , Little Rock, AR, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT03733041/ICF_000.pdf